CLINICAL TRIAL: NCT00393705
Title: A Comparison of Insulin Lispro MM Intensive Mixture Therapy With Progressive Dose-Titration of Insulin Lispro LM or Biphasic Insulin Aspart 30/70
Brief Title: Lispro Mid Mixture (MM) Intensive Mixture Therapy With Progressive Dose-Titration of Lispro Low Mixture (LM) or Biphasic Insulin Aspart 30/70 (S019)
Acronym: S019
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10916; F3Z-VI-S019 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Results first posted 2010-04-27 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin lispro LM + insulin lispro MM (Experimental): Three times per day subcutaneous injection of insulin lispro mid mixture (MM) with the possibility to change the evening injection of MM to insulin lispro low mixture (LM) if fasting blood glucose target is not achieved.
  Interventions: Drug: insulin lispro LM; Drug: insulin lispro MM
- Insulin Biphasic Aspart 30/70 or Insulin Lispro LM (Active Comparator): Twice daily subcutaneous injection of either insulin biphasic aspart 30/70 or insulin lispro low mixture (LM) (continuation of analogue formulation used before study enrollment).
  Interventions: Drug: Insulin Biphasic Aspart 30/70; Drug: insulin lispro LM

INTERVENTIONS:
Drug: Insulin Biphasic Aspart 30/70 — Participant adjusted dose, twice daily, injected subcutaneously for 16 weeks
  Arms: Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Drug: insulin lispro LM — Participant adjusted dose, injected subcutaneously for 16 weeks - possibility of using instead of insulin lispro MM before evening meal if there is a risk of hypoglycemia after the dinner or high fasting glucose levels.
  Other Names: Low Mix; Humalog
  Arms: insulin lispro LM + insulin lispro MM
Drug: insulin lispro MM — Participant adjusted dose, three times per day, injected subcutaneously for 16 weeks
  Other Names: Mid Mix; Humalog
  Arms: insulin lispro LM + insulin lispro MM
Drug: insulin lispro LM — Participant adjusted dose, twice daily, injected subcutaneously for 16 weeks
  Other Names: Low Mix; Humalog
  Arms: Insulin Biphasic Aspart 30/70 or Insulin Lispro LM

SUMMARY:
Investigation into patients with type 2 diabetes mellitus not achieving adequate glycemic control while treated with combination of premixed insulin analogue formulations twice daily and metformin will be randomly assigned to follow one of two insulin treatment strategies used in combination with metformin administration. The aim of the trial is to try to achieve optimal metabolic control and explore full therapeutic potential of the strategies, patients in both arms will follow progressive insulin dose titration algorithms for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes (World Health Organization [WHO] classification).
* Are at least 30 years of age and less than 75 years of age.
* Have been receiving hypoglycemic treatment with premixed insulin analogue (either with insulin lispro LM or biphasic insulin aspart 30/70) administered twice daily in combination with at least 1500 milligrams (mg) of metformin per day for at least 60 days immediately prior to the study.
* Have a hemoglobin A1c 1.2 to 1.8 times the upper limit of the normal reference range at the local laboratory at Visit 1 or
* Have at least 6 of 9 of the postprandial blood glucose values recorded in the period between Visit 1 and Visit 2 exceeding 180 milligrams per 100 milliliters (mg/dl) (10.0 millimole per liter [mmol/l]).
* Have given written informed consent to participate in this study in accordance with local regulations.

Exclusion Criteria:

* Are taking any other oral anti-diabetic medication (OAM) not mentioned in inclusion criterion.
* Have a body mass index greater than 40 kilograms per meter squared (kg/m2).
* Have had more than one episode of severe hypoglycemia within 6 months prior to entry into the study.
* Have congestive heart failure.
* Have an irregular sleep/wake cycle (for example, patients who sleep during the day and work during the night).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2006-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb, Croatia
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rzeszów
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest, Romania
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kempton Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kenilworth
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuilsriver
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Konya

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Lispro LM + Insulin Lispro MM: Three times per day insulin lispro mid mixture (MM) with the possiblity to change the evening injection of MM to insulin lispro low mixture (LM) if fasting blood glucose target is not achieved.
  Insulin lispro mid mixture (MM): Participant adjusted dose, three times per day, injected subcutaneously for 16 weeks.
  Insulin lispro low mixture (LM): Participant adjusted dose, possibly in the evening.
- Insulin Biphasic Aspart 30/70 or Insulin Lispro LM: Twice daily treatment of either biphasic insulin aspart 30/70 or insulin lispro LM (continuation of analogue formulation used before study enrollment).
  Insulin Biphasic Aspart 30/70: Participant adjusted dose, twice daily, injected subcutaneously for 16 weeks.
  Insulin Lispro LM: Participant adjusted dose, twice daily, injected subcutaneously for 16 weeks.
Period: Overall Study
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Started | 151 | 151
Received at Least One Dose of Study Drug | 139 | 139
Completed | 128 | 128
Not Completed | 23 | 23
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Entry Criteria Not Met | 10 | 10
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM | Total
Number analyzed (Participants) | 151 | 151 | 302
Age Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.50) | 58.4 (9.01) | 57.7 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 82 | 174
  Male | 59 | 69 | 128
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 150 | 149 | 299
  African | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Poland | 33 | 33 | 66
  Croatia | 7 | 11 | 18
  Turkey | 33 | 45 | 78
  Romania | 37 | 28 | 65
  South Africa | 12 | 13 | 25
  Hungary | 29 | 21 | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 32.3 (4.11) | 31.0 (4.27) | 31.7 (4.23)
Daily Dose of Antihyperglycaemic Therapy Prior to Study (International Units [IU]) [Mean (Standard Deviation); unit: International Units (IU)]
  Insulin Lispro Dose (n=61, n=57) | 45.8 (16.87) | 39.7 (13.79) | 42.9 (15.69)
  Biphasic Insulin Aspart 30/70 Dose (n=90, n=94) | 47.5 (20.31) | 44.0 (17.79) | 45.7 (19.09)
Daily Dose of Metformin Treatment Prior to Study (milligrams [mg]) [Mean (Standard Deviation); unit: milligrams (mg)] | 1898.8 (402.99) | 1863.9 (379.00) | 1881.4 (390.92)
Duration of Antihyperglycaemic Therapy Prior to Study [Mean (Standard Deviation); unit: months]
  Insulin Treatment | 42.8 (41.65) | 43.7 (51.50) | 43.3 (46.76)
  Premixed Insulin Analogue Treatment | 16.4 (17.61) | 16.1 (22.42) | 16.3 (20.12)
  Oral Hypoglycemic Treatment | 54.7 (56.55) | 58.9 (64.56) | 56.8 (60.62)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 10.9 (5.66) | 11.5 (7.19) | 11.2 (6.47)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 182.6 (46.15) | 185.4 (59.22) | 184.0 (53.04)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 165.4 (9.47) | 165.4 (9.82) | 165.4 (9.63)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c] | 8.6 (1.27) | 8.5 (1.20) | 8.5 (1.23)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 88.6 (14.97) | 85.1 (14.45) | 86.8 (14.79)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) at 16 Week Endpoint
Time Frame: 16 weeks
Population: Number of patients who received at least one dose of study drug and had an HbA1c measure at endpoint.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 131 | 135
percent HbA1c | 7.71 (1.098) | 7.84 (1.036)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.2519, ANCOVA; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

2. Secondary Outcome: Percentage of Patients Achieving Hemoglobin A1c (HbA1c) <7% and HbA1c ≤6.5% at 16 Week Endpoint
Time Frame: 16 weeks
Population: Number of patients who received at least one dose of study drug and had a post-baseline HbA1c value at endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 131 | 135
percentage of participants
  HbA1c <7% | 21.4 | 18.5
  HbA1c ≤6.5% | 11.5 | 6.7
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0287, Regression, Logistic — P-value for HbA1c <7%. Additional statistically significant terms from the model below were baseline HbA1c and treatment by lead-in interaction; Model: Logit(p(response)/1-p(response)) = U + r' X, where u = intercept parameter, X = vector of parameters (treatment, baseline value, lead-in)
Statistical Analysis 2: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0471, Regression, Logistic — P-value for HbA1c ≤6.5%. Additional statistically significant term from the model below was baseline HbA1c; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at 16 Week Endpoint
Time Frame: Baseline, 16 Weeks
Population: Number of patients who received at least one dose of study drug and a post-baseline HbA1c value at endpoint.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 131 | 135
percent HbA1c | -1.00 (1.019) | -0.82 (0.970)

4. Secondary Outcome: 2-hour Postprandial Plasma Glucose Concentrations After the Midday Meal From Self-monitored 7-point Plasma Glucose at 16 Week Endpoint
Description: Participants self-monitored their blood glucose concentrations at 7 time points: three premeal and three 2-hour postprandial meal measurements for the morning (breakfast), midday (lunch), and evening (dinner) meals, as well as a 3:00 AM measurement. Results presented here are for the blood glucose concentrations 2-hours after the midday meal at Week 16.
Time Frame: 16 weeks
Population: Number of patients who received at least one dose of study drug and had a post-baseline 2-hour postprandial plasma glucose reading after the midday meal at week 16.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 125 | 126
milligrams per deciliter (mg/dL) | 163.4 (40.85) | 178.2 (48.54)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0077, ANCOVA; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

5. Secondary Outcome: Mean 2-hour Postprandial Blood Glucose Excursions After Midday Meal at 16 Week Endpoint
Description: Participants self-monitored their blood glucose concentrations at 7 time points: three premeal and three 2-hour postprandial meal measurements for the morning (breakfast), midday (lunch), and evening (dinner) meals, as well as a 3:00 AM measurement. Results presented here are for the difference (excursion) between midday premeal and 2-hour postprandial midday meal blood glucose concentrations at Week 16.
Time Frame: 16 weeks
Population: Number of patients who received at least one dose of study drug and had a post-baseline 2-hour postprandial blood glucose reading after the midday meal at week 16.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 125 | 127
milligrams per deciliter (mg/dL) | 17.0 (36.42) | 36.1 (48.20)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0002, ANCOVA; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

6. Secondary Outcome: Mean Daily Blood Glucose Values at 16 Week Endpoint
Time Frame: 16 weeks
Population: Number of patients who received at least one dose of study drug and had a post-baseline blood glucose reading at week 16 for the respective variable.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 125 | 127
milligrams per deciliter (mg/dL)
  Fasting | 161.1 (35.41) | 153.9 (35.84)
  2-Hours After Breakfast | 179.0 (46.14) | 160.9 (45.25)
  Pre-Lunch | 146.3 (34.75) | 141.7 (41.72)
  2-Hours After Lunch | 163.4 (40.85) | 178.2 (48.54)
  Pre-Dinner | 157.5 (41.28) | 165.7 (47.77)
  2-Hours After Dinner | 166.4 (44.13) | 171.4 (45.92)
  3:00 A.M. | 141.2 (32.19) | 141.0 (35.08)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0129, ANCOVA — P-value for Fasting; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 2: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0027, ANCOVA — P-value for 2-Hours After Breakfast; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 3: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.1947, ANCOVA — P-value for Pre-Lunch; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 4: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0077, ANCOVA — P-value for 2-Hours After Lunch; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 5: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.1885, ANCOVA — P-value for Pre-Dinner; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 6: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.5525, ANCOVA — P-value for 2-Hours After Dinner; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 7: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.4994, ANCOVA — P-value for 3:00 A.M; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

7. Secondary Outcome: Number of Patients With Self-reported Hypoglycemic Episodes
Description: Hypoglycemia: any time a patient feels, or another person observes, that patient is experiencing a sign/symptom that he or she would associate with hypoglycemia or a plasma-equivalent glucose measurement ≤70 mg/dL. Nocturnal hypoglycemia: hypoglycemia occurring after bedtime and prior to morning meal and morning dose of insulin or metformin. Severe hypoglycemia: hypoglycemia where patient requires assistance from another person and which is associated with either a blood glucose level less than 50 mg/dL or prompt recovery after oral carbohydrate, intravenous glucose or glucagon administration.
Time Frame: Baseline through 16 weeks
Population: Number of patients who received at least one dose of study drug and had at least one assessment after randomization.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 139 | 139
participants
  1 Hypoglycemic Event | 24 | 14
  2 Hypoglycemic Events | 9 | 11
  ≥3 Hypoglycemic Events | 24 | 33
  1 Nocturnal Hypoglycemic Event | 10 | 14
  2 Nocturnal Hypoglycemic Events | 3 | 3
  ≥3 Nocturnal Hypoglycemic Events | 2 | 8
  1 Severe Hypoglycemic Event | 1 | 0
  2 Severe Hypoglycemic Events | 1 | 1

8. Secondary Outcome: 30-Day Adjusted Rate of Hypoglycemic Events
Description: as for outcome 7
Time Frame: Baseline through 16 weeks
Population: Number of patients who received at least one dose of study drug and had at least one assessment after randomization.
Measure: Mean (Standard Deviation); unit: number of events per 30 days
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 139 | 139
number of events per 30 days
  Total Hypoglycemic Episodes/30 Days | 0.52 (1.212) | 0.64 (1.398)
  Nocturnal Hypoglycemic Episodes/30 Days | 0.04 (0.138) | 0.12 (0.361)
  Severe Hypoglycemic Episodes/30 Days | 0.01 (0.046) | 0 (0.045)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.7230, ANCOVA — P-value for Total Hypoglycemic Episodes/30 Days; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 2: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0063, ANCOVA — P-value for Nocturnal Hypoglycemic Episodes/30 Days; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 3: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.8876, ANCOVA — P-value for Severe Hypoglycemic Episodes/30 Days; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

9. Secondary Outcome: Change From Baseline in Weight at 16 Week Endpoint
Time Frame: Baseline, 16 weeks
Population: Number of patients who received at least one dose of study drug and had at least one post-baseline weight value at week 16.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 126 | 127
kilograms (kg) | 1.3 (2.73) | 0.4 (2.45)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0009, ANCOVA; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

10. Secondary Outcome: Total Daily Insulin Dose at 4 Weeks and 12 Weeks
Time Frame: 4 weeks and 12 weeks
Population: Number of patients who received at least one dose of study drug and had a post-baseline insulin measurement at week 4 and week 12.
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Number analyzed (Participants) | 134 | 135
International Units (IU)
  4 Weeks (n=134, n=135) | 57.1 (22.32) | 51.4 (18.90)
  12 Weeks (n=130, n=131) | 64.4 (25.63) | 58.0 (22.90)
Statistical Analysis 1: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0056, ANCOVA — P-value for Week 4; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error
Statistical Analysis 2: Comparison: Insulin Lispro LM + Insulin Lispro MM vs Insulin Biphasic Aspart 30/70 or Insulin Lispro LM; Test type: Superiority or Other; p = 0.0421, ANCOVA — P-value for Week 12; Model: Value = Treatment + Lead-in + Treatment*Lead-in + Visit + Treatment*Visit + Value at baseline + error

ADVERSE EVENTS:
Arm/Group | Insulin Lispro LM + Insulin Lispro MM | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM
Serious Adverse Events (participants affected / at risk) | 3/139 | 7/139
Other Adverse Events (participants affected / at risk) | 26/139 | 26/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro LM + Insulin Lispro MM (N=139) | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM (N=139)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) — One myocardial infarction resulted in death during the study. However, another patient had a fatal myocardial infarction after study completion but within the 30 day follow-up window for adverse events after completion.
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro LM + Insulin Lispro MM (N=139) | Insulin Biphasic Aspart 30/70 or Insulin Lispro LM (N=139)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 2 (3)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 7 (8)
Oral herpes (Infections and infestations) | 0 (0) | 1 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Dental care (Surgical and medical procedures) | 1 (1) | 0 (0)
Eye laser surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Influenza immunisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days